CLINICAL TRIAL: NCT00872027
Title: Feasibility Study to Prevent Post-ICU Depression
Brief Title: Preventing Depression in People Receiving Mechanical Ventilation in an Intensive Care Unit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R34MH082156 (NIH); R34MH082156 (NIH); DSIR 83 ATP
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Depression
Keywords: Critical Illness; Intensive Care Unit; Acute Respiratory Failure; Prolonged Mechanical Ventilation
MeSH Terms: conditions — Depression; Critical Illness | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive 8 weeks of escitalopram treatment.
  Interventions: Drug: Escitalopram
- 2 (Placebo Comparator): Participants will receive 8 weeks of placebo pills.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — 10 mg of escitalopram administered enterally with the option for dose escalation to 20 mg after 3 to 5 weeks if the medical condition is stable and no liver disease presents
  Other Names: Lexapro
  Arms: 1
Drug: Placebo — Placebo pills for 8 weeks
  Arms: 2

SUMMARY:
This study will determine the effectiveness of antidepressant medication in preventing depression and improving recovery in people who have been supported by mechanical ventilators in an intensive care unit (ICU).

DETAILED DESCRIPTION:
More than one third of all people admitted to ICUs in hospitals require mechanical ventilation for respiratory failure. Many people who survive after being on mechanical ventilation for a prolonged time have significant issues with recovery and quality of life when discharged from the ICU. They are also more prone to depression, which increases patient suffering and the need for medical care, decreases quality of life, and is associated with increased mortality. Previous research indicates that antidepressant medications may improve quality of life and recovery in people who have had a heart attack, but that behavioral treatments are not effective in this case. Treating depression in ICU patients with respiratory failure has not been examined. In this study, antidepressant medications will be given to people who have been on mechanical ventilation in an ICU to determine the effectiveness of antidepressants in improving medical recovery and quality of life. Only a small number of participants will be enrolled in this trial to test the methods and theory; if it is successful, a larger trial will be conducted to determine whether these findings can be widely generalized.

Participation in this study will last 8 weeks, with follow-up assessments lasting for 6 months. Participants on a ventilation machine will be randomly assigned to receive either escitalopram, which is an FDA-approved antidepressant, or a placebo pill. A healthy surrogate may need to enroll participants in the study, because participants will begin treatment while in the ICU and may not be able to make an informed decision. The medication or placebo treatment will last for 2 months, continuing at the participant's home after discharge from the ICU. Dosage levels will begin at 10 mg per day and will be increased to 20 mg per day for some participants after 3 to 5 weeks. Every 2 weeks, participants will complete questionnaires by phone or in person about their medical and psychological symptoms and about whether they are taking the study medication. At 8 weeks, participants will complete an in-person interview about depression symptoms, quality of life, and physical function. At 9 weeks, participants will complete a telephone interview about medication withdrawal. Finally, at 4 and 6 months, participants will complete interviews about depression and general health.

ELIGIBILITY:
Inclusion Criteria:

* Newly mechanically ventilated via an endotracheal tube
* Expected to remain intubated for at least 48 hours
* Fluent in English or Spanish

Exclusion Criteria:

* Depression before admission to the ICU, as determined by a proxy interview
* Use of antidepressant medication within the last 2 weeks or a monoamine oxidase (MAO) inhibitor in the previous month
* History of suicide attempt
* Ventricular arrhythmias or a seizure requiring medication in the last 6 months
* History of retinal vascular proliferation or bleeding
* Migraine headaches treated with 5-HT1 agonists
* Organ transplant within the last 6 months
* Score of less than 4 on the Glasgow coma scale, in the absence of drug effects, for 2 days
* Acute brain hemorrhage
* Increased intracranial pressure
* Active bleeding or less than 20,000 platelets/ul
* Expected prolonged inability to enterally administer escitalopram
* Residence more than 75 miles from study facility
* Serum sodium less than 125 mEq/l
* Hypersensitivity to citalopram or escitalopram
* Pregnant, breastfeeding, or possibly becoming pregnant in the next 3 months
* Undergoing life-support withdrawal or very low likelihood of 2-month survival
* Cognitive or communication impairment severe enough to preclude a conversation with an interviewer present before admission to ICU

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Weinert, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Will Receive 8 Weeks of Escitalopram Treatment.: Participants will receive 8 weeks of escitalopram treatment.
  Escitalopram: 10 mg of escitalopram administered enterally with the option for dose escalation to 20 mg after 3 to 5 weeks if the medical condition is stable and no liver disease presents
- Participants Will Receive 8 Weeks of Placebo Pills.: Participants will receive 8 weeks of placebo pills.
  Placebo: Placebo pills for 8 weeks
Period: Overall Study
Arm/Group | Participants Will Receive 8 Weeks of Escitalopram Treatment. | Participants Will Receive 8 Weeks of Placebo Pills.
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Will Receive 8 Weeks of Escitalopram Treatment. | Participants Will Receive 8 Weeks of Placebo Pills. | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 7 | 8 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility, Defined as the Number of Participants Recruited and Administered a Medication Dose Within 48 Hours of Mechanical Ventilation
Time Frame: Measured within 2 days of participant recruitment
Measure: Number; unit: participants
Arm/Group | Participants Will Receive 8 Weeks of Escitalopram Treatment. | Participants Will Receive 8 Weeks of Placebo Pills.
Number analyzed (Participants) | 7 | 8
participants | 7 | 8

ADVERSE EVENTS:
Time Frame: These were collected over a 48 hour period.
Description: Adverse event collection was done by body system and not specific event.
Arm/Group | Participants Will Receive 8 Weeks of Escitalopram Treatment. | Participants Will Receive 8 Weeks of Placebo Pills.
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Will Receive 8 Weeks of Escitalopram Treatment. (N=7) | Participants Will Receive 8 Weeks of Placebo Pills. (N=8)
GI (Gastrointestinal disorders) | 5 (5) | 7 (7)
Heart (Cardiac disorders) | 1 (4) | 4 (4)
Skin (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (4)
Nervous Sytem (Nervous system disorders) | 1 (3) | 2 (3)
Eye/Ear (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Genital/Urinary (Renal and urinary disorders) | 2 (4) | 4 (4)
Sleep (General disorders) | 2 (5) | 3 (4)
Other (General disorders) | 3 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No